Official Title: Effects of 20 Minutes Osteoporosis Education on the Awareness of Osteoporosis in People Registered in Elderly Care Homes.

NCT05936177

Date of the Document: June 8, 2023

## **Informed Consent Form**

Osteoporosis is a disease that poses a threat to the elderly population. This study is designed to assess the osteoporosis awareness of individuals at risk. Volunteers will be asked to complete a questionnaire for this purpose.

Those who complete the questionnaire may, if they wish, attend an education session on 'Osteoporosis' to be held at the Elderly House under the auspices of the Muratpaşa Municipality. The education will be conducted by a Physical Medicine and Rehabilitation physician, who will deliver a 20-minute presentation containing verbal and visual information about osteoporosis, prevention methods, and treatments.

The presentation will provide you with knowledge about osteoporosis, preventive measures, familiarity with proper nutrition and exercise content. This information will offer you options for prevention against future hip fractures, spinal fractures, pain, and mobility difficulties.

Participants attending the presentation can ask questions and seek assistance from the Physical Medicine physician regarding this topic.

Volunteers who participate in the presentation can fill out a short questionnaire immediately after the presentation and again 1 month later. The time spent filling out the questionnaire is approximately 5 minutes, and if you choose to attend the presentation, it will take about 20 minutes. You are free to discontinue your participation at any stage of the research. Forms containing name and phone number information will be kept confidential, and even if the research results are published, they will not contain any personal identifying information. There is no cost associated with the research, and no burden will be placed on you or your social security institution.

For any questions related to the research or your rights, you can contact the following person and phone number, available 24 hours a day: Dr. Selkin Yılmaz Muluk ...

You are participating in this study voluntarily. You have the right to refuse to participate in the research. If you decide not to continue after the research has started, you still have this right. Even if you choose not to participate in the study, you may still listen to the presentation.

'I have read the information that should be given to the volunteer before the research. These were explained to me in writing and verbally. With my own consent, without any pressure or coercion, I agree to participate in this research.'

I have read the above information. I understand the necessary explanations provided by the doctor. I agree to participate in this study of my own free will.

Name and Signature of Volunteer: Name and Signature of Researcher Providing

Explanations: Name, Signature, and Position of Witness throughout the Consent Process